CLINICAL TRIAL: NCT03570645
Title: Comparison of the Duration of Ropivacaine Combined With Dexmedetomidine or Dexamethasone on Paravertebral Block in Patients Undergoing Video-assisted Thoracic Surgery
Brief Title: Comparison of the Duration of Ropivacaine Combined With Dexmedetomidine or Dexamethasone on Paravertebral Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Wen-fei Tan, Professor, China Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20180616
Record Dates: First submitted 2018-06-16; First posted 2018-06-27 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: thoracic paravertebral blocks using a combination of ropivacaine and dexmedetomidine or dexamethasone
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- dexmedetomidine group (Experimental): thoracic paravertebral blocks using a combination of ropivacaine and dexmedetomidine 100 ug every time
  Interventions: Drug: Dexmedetomidine Group
- dexamethasone Group (Experimental): thoracic paravertebral blocks using a combination of ropivacaine and dexamethasone 10 mg every time
  Interventions: Drug: dexamethasone group
- control group (Sham Comparator): thoracic paravertebral blocks using only ropivacaine
  Interventions: Drug: control group

INTERVENTIONS:
Drug: Dexmedetomidine Group — combination of ropivacaine and dexmedetomidine 100 ug every time
  Arms: dexmedetomidine group
Drug: dexamethasone group — combination of ropivacaine and dexamethasone 10mg every time
  Arms: dexamethasone Group
Drug: control group — block with only ropivacaine
  Arms: control group

SUMMARY:
This study was a prospective, randomized, controlled, and double-blind trial. Major assessments were made during the operation and 48 h postoperatively.

DETAILED DESCRIPTION:
The prime outcomes were the time in minutes from leave the postoperative care unit to the first patient-controlled intravenous analgesia press.The secondary outcomes were to compare the following: (1)blood concentrations of ropivacaine was measured at 0.5 h, 1 h, 2 h, 3 h, and 24 h after paravertebral nerve block; and (2) the patient's intraoperative opioid use, phenylephrine use, fluid intake, urine output, dry mouth score, and 24 h and 48 h visual analogue scale.

ELIGIBILITY:
Inclusion Criteria:

* (1) age 18 to 65 years,
* (2) scheduled to undergo video-assisted thoracic surgery,
* (3) American Society of Anesthesiologists risk classification I-II.

Exclusion Criteria:

* (1) patient refusal;
* (2) known hypersensitivity to the study medication (ropivacaine);
* (3) long-term use of opioids;
* (4) liver or renal insufficiency;
* (5) a history of psychiatric or neurological disease;
* (6) deafness;
* (7) regular use of acetaminophen, nonsteroidal anti-inflammatory drugs, corticosteroids, or antiemetics; and
* (8) a preoperative Pittsburgh Sleep Quality Index (PSQI) global score higher than 6.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-18 (Actual)

PRIMARY OUTCOMES:
Change of thoracic paravertebral block analgesia duration | Change from Baseline to 2 days after surgery
  The prime outcomes were the time in minutes from leave the postoperative care unit to the first patient-controlled intravenous analgesia press

SECONDARY OUTCOMES:
blood concentrations of ropivacaine | Change from Baseline to 2 days after surgery
  (The secondary outcomes were to compare the following: (1)blood concentrations of ropivacaine was measured at 0.5 h, 1 h, 2 h, 3 h, and 24 h after paravertebral nerve block; and (2) the patient's intraoperative opioid use, phenylephrine use, fluid intake, urine output, dry mouth score, and 24 h and 48 h visual analogue scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, the First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided